CLINICAL TRIAL: NCT04941105
Title: Impact of PCSK9 Inhibition on Clinical Outcome in Patients During the Inflammatory Stage of the COVID-19: the Randomized, Double-blind, Phase III IMPACT-SIRIO 5 Study.
Brief Title: Impact of PCSK9 Inhibition on Clinical Outcome in Patients During the Inflammatory Stage of the COVID-19
Acronym: IMPACT-SIRIO 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Head of Department of Cardiology and Internal Medicine, Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMPACT-SIRIO 5
Record Dates: First submitted 2021-06-21; First posted 2021-06-28 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Sars-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2 Pneumonia; PCSK9 inhibitor
MeSH Terms: conditions — COVID-19 | interventions — evolocumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCSK9 inhibitor (evolocumab) (Experimental): 140 mg of evolocumab as a single subcutaneous injection and standard of care accordance to the latest recommendations
  Interventions: Drug: Evolocumab
- Usual Care (Placebo Comparator): 1 ml of 0,9% saline solution as a single subcutaneous injection. Patients will be treated in accordance to the latest recommendations on caring for patients infected with SARS-CoV-2.
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Evolocumab — A single subcutaneous administration of 140 mg evolocumab
  Arms: PCSK9 inhibitor (evolocumab)
Drug: Saline solution — A single subcutaneous injection of 1ml of 0,9% saline solution
  Arms: Usual Care

SUMMARY:
The IMPACT-SIRIO 5 is a randomized, double-blind, phase III clinical trial aimed to evaluate safety and efficacy of PCSK9 inhibition on clinical outcome in patients during the inflammatory stage of the COVID-19. During the hospitalization participants will be randomized in a 1:1 ratio to either receive PCSK9 inhibitor (evolocumab) or to receive placebo (saline solution). Furthermore, all people included in the study will be treated in accordance to the latest recommendations on the treatment of patients infected with SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for participation in the study
2. Male and female age 18 or more at the time of signing the informed consent
3. SARS-CoV-2 infection confirmed by Real-Time Reverse Transcription Polymerase Chain Reaction (RT-PCR)
4. COVID-19 pneumonia with a typical radiological changes
5. PaO2/FIO2 ratio less than or equal to 300
6. COVID-19 Pneumonia in cytokine storm with elevated serum level of interleukin-6

Exclusion Criteria:

1. Use of fibrates other than fenofibrate or fenofibric acid
2. Known active infections or other clinical condition that contraindicate PCSK9 inhibitors
3. Known systemic hypersensitivity to PCSK9 inhibitors
4. Estimated glomerular filtration rate <30 ml/min/1.73 m2
5. Absolute neutrophil count (ANC) less than 2000/mm3
6. A platelet count less than 50000/mm3
7. Creatine kinase (CK) greater than 3x upper limit of normal (ULN)
8. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 3x upper limit of normal (ULN)
9. Not expected to survive for more than 48 hours from screening
10. Unrelated co-morbidity with life expectancy <3 months.
11. Pregnancy
12. Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient by their participation in the study
13. Patient being treated with other immunomodulators (except for glucocorticoids).
14. Patient included in any other interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Death from any cause or need for intubation | during hospitalization, up to 30 days
  Indication for intubation determined individually for each patient and clinical status

SECONDARY OUTCOMES:
Change in serum interleukin-6 concentration from day 0 to day 7 and day 30 | 7 and 30 days from randomization
Death from any cause | during hospitalization, up to 30 days
  Death from any cause during hospitalization.
Need for intubation | during hospitalization, up to 30 days
  Indication for intubation determined individually for each patient and clinical status
Duration of oxygen therapy | during hospitalization, up to 30 days
  Defined as the number of days of oxygen therapy (including all methods of oxygen therapy)
Duration of hospital stay | during hospitalization, up to 30 days
  Defined as the number of days that pass between the day of hospital admission and discharge or death.
Days of intubation | during hospitalization, up to 30 days
  Defined as the number of days between intubation and extubation
Time with Non-invasive mechanical ventilation (NIV) or High-flow nasal cannula (HFNC) | during hospitalization, up to 30 days
  Defined as the number of days between initiation and cessation of Non-invasive mechanical ventilation (NIV) or High-flow nasal cannula (HFNC)

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, MD, PhD, Principal Investigator — Collegium Medicum, Nicolaus Copernicus University, Bydgoszcz, Poland; Eliano Navarese, Md, PhD, Principal Investigator — Collegium Medicum, Nicolaus Copernicus University, Bydgoszcz, Poland
Locations (1):
- Antoni Jurasz University Hospital No. 1, Bydgoszcz, Poland

REFERENCES:
- [Derived] Navarese EP, Podhajski P, Gurbel PA, Grzelakowska K, Ruscio E, Tantry U, Magielski P, Kubica A, Niezgoda P, Adamski P, Junik R, Przybylski G, Pilaczynska-Cemel M, Rupji M, Specchia G, Pinkas J, Gajda R, Gorog DA, Andreotti F, Kubica J. PCSK9 Inhibition During the Inflammatory Stage of SARS-CoV-2 Infection. J Am Coll Cardiol. 2023 Jan 24;81(3):224-234. doi: 10.1016/j.jacc.2022.10.030. PMID 36653090